CLINICAL TRIAL: NCT06863545
Title: Further Lipid-Lowering With PCSK9 Inhibitors for Cardiovascular Outcomes in High-Risk Coronary Plaques Assessed by CT Angiography
Acronym: FLAVOUR IV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0052
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease; CT Angiography; PCSK9; Cardiovascular Events
Keywords: PCSK9 inhibitors; Lipid-lowering therapy; High-Risk Coronary Plaques; Coronary CT angiography
MeSH Terms: conditions — Coronary Artery Disease | interventions — PCSK9 Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCSK9 inhibitors plus background lipid-modifying therapy (Experimental): Patients will receive PCSK9 inhibitors treatment and background lipid-modifying therapy for the first 12 months after randomization, and then continue background lipid-modifying therapy for the remainder of the trial.
- Standard lipid-modifying therapy (Active Comparator): Patients will receive standard LMT commonly used in clinical practice.
  Interventions: Drug: Standard lipid-modifying therapy

INTERVENTIONS:
Drug: PCSK9 inhibitors and background lipid-modifying therapy — Patients will receive subcutaneous injections of PCSK9 inhibitors and oral administration of background LMT (including statins and/or cholesterol absorption inhibitors) for the first 12 months after randomization, with PCSK9 inhibitors administered every 2 weeks. After the first 12 months, patients will discontinue the PCSK9 inhibitors but continue background LMT for the remainder of the trial.
Drug: Standard lipid-modifying therapy — Patients will receive standard LMT commonly used in clinical practice.
  Arms: Standard lipid-modifying therapy

SUMMARY:
The primary objective was to evaluate the effect of PCSK9 inhibitors in addition to the background lipid-modifying therapy (LMT), compared with standard LMT in terms of clinical outcomes in patients with coronary CT angiography (CCTA)-detected high-risk plaques.

DETAILED DESCRIPTION:
CCTA is an accurate, noninvasive alternative to invasive coronary angiography. CCTA can provide detailed information about the characteristics of coronary artery plaques, such as their composition, morphology, and distribution. Various CCTA-detected plaque characteristics indicative of plaque quantity and quality have been identified as high-risk features independently predicting clinical events, including the presence of positive remodeling, low attenuation plaque, spotty calcification, and napkin ring sign. Currently, the treatment for CCTA-detected high-risk plaque has been receiving increasing interest. The current study aimed to prove the efficacy of PCSK9 inhibitors in addition to the background LMT, as compared with standard LMT in patients with CCTA-detected high-risk plaques.

Hypothesis: PCSK9 inhibitors in addition to background LMT will show a superior event rate, compared with standard LMT, in terms of major adverse cardiac and cerebrovascular events (MACCEs) at 24 months after the last patient's randomization in patients with high-risk coronary plaques assessed by CT Angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years.
2. Patients with at least one target lesion meet CCTA-detected plaque features of the following:

   1. Degree of stenosis ≥ 50% or plaque burden ≥ 70%
   2. At least 2 of the following high-risk plaque features:

   i. Low-attenuation plaque ii. Positive remodeling iii. Napkin-ring sign iv. Spotty calcium
3. The target lesion is located at the proximal or mid segment of left anterior descending artery, left circumflex artery or right coronary artery.
4. Subject is able to confirm his/her understanding of the risks, benefits, and treatment alternatives of receiving study-related treatment. He/she or his/her legally authorized representative provides written informed consent prior to any study-related procedure.

Exclusion Criteria:

1. Target lesions underwent or planned to revascularization.
2. Patients with acute coronary syndrome.
3. New York Heart Association class III or IV, or last known left ventricular ejection fraction < 30%.
4. Uncontrolled or recurrent ventricular tachycardia.
5. Homozygous familial hypercholesterolemia.
6. Active liver disease or hepatic dysfunction.
7. Failed CCTA plaque analysis.
8. Non-cardiac co-morbid conditions with life expectancy < 2 years.
9. Pregnant and/or lactating women.
10. Known hypersensitivity or contraindication to statin or PCSK9 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3596 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCEs) | 24 months after the last patient's randomization
  A composite of death from any cause, myocardial infarction (MI), coronary revascularization, or stroke.

SECONDARY OUTCOMES:
MACCEs | 60 months after the last patient's randomization
  a composite of death from any cause, MI, coronary revascularization, or stroke.
Individual component of MACCEs. | 24 and 60 months after the last patient's randomization
  Individual component of MACCEs (death from any cause, MI, coronary revascularization, or stroke)
Major adverse cardiovascular events (MACEs) | 24 and 60 months after the last patient's randomization
  Defined as a composite of death from any cause, MI, coronary revascularization.
Target vessel failure (TVF) | 24 and 60 months after the last patient's randomization
  Defined as a composite of cardiac death, target-vessel MI, or target vessel revascularization
Cost-effectiveness analysis | 24 and 60 months after the last patient's randomization
  Cost-effectiveness analysis
All-cause and cardiac death. | 24 and 60 months after the last patient's randomization
  All-cause and cardiac death.
Any target-vessel MI. | 24 and 60 months after the last patient's randomization
  Any target-vessel MI.
Any target vessel revascularization. | 24 and 60 months after the last patient's randomization
  Any target vessel revascularization.
Any coronary revascularization (ischemia-driven or all). | 24 and 60 months after the last patient's randomization
  Any coronary revascularization (ischemia-driven or all).
CT coronary angiography findings | 36 months after the last patient's randomization
  Changes in the CT-derived fractional flow reserve, lumen, plaque quantity and quality between baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyang Hu, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Bon-Kwon Koo, Principal Investigator — Seoul National University Hospital
Locations (6):
- China (5):
  - Zhejiang Provincial Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - Hangzhou Linping First People's Hospital, Hangzhou
  - The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - Jinhua Central Hospital, Jinhua
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The deidentified data will be shared after publication of first manuscript.
Supporting Information: Study Protocol
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Iatan I, Guan M, Humphries KH, Yeoh E, Mancini GBJ. Atherosclerotic Coronary Plaque Regression and Risk of Adverse Cardiovascular Events: A Systematic Review and Updated Meta-Regression Analysis. JAMA Cardiol. 2023 Oct 1;8(10):937-945. doi: 10.1001/jamacardio.2023.2731. PMID 37647074
- [Background] Nicholls SJ, Puri R, Anderson T, Ballantyne CM, Cho L, Kastelein JJ, Koenig W, Somaratne R, Kassahun H, Yang J, Wasserman SM, Scott R, Ungi I, Podolec J, Ophuis AO, Cornel JH, Borgman M, Brennan DM, Nissen SE. Effect of Evolocumab on Progression of Coronary Disease in Statin-Treated Patients: The GLAGOV Randomized Clinical Trial. JAMA. 2016 Dec 13;316(22):2373-2384. doi: 10.1001/jama.2016.16951. PMID 27846344
- [Background] Raber L, Ueki Y, Otsuka T, Losdat S, Haner JD, Lonborg J, Fahrni G, Iglesias JF, van Geuns RJ, Ondracek AS, Radu Juul Jensen MD, Zanchin C, Stortecky S, Spirk D, Siontis GCM, Saleh L, Matter CM, Daemen J, Mach F, Heg D, Windecker S, Engstrom T, Lang IM, Koskinas KC; PACMAN-AMI collaborators. Effect of Alirocumab Added to High-Intensity Statin Therapy on Coronary Atherosclerosis in Patients With Acute Myocardial Infarction: The PACMAN-AMI Randomized Clinical Trial. JAMA. 2022 May 10;327(18):1771-1781. doi: 10.1001/jama.2022.5218. PMID 35368058
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Schwartz GG, Steg PG, Szarek M, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Pordy R, Quintero K, Roe MT, Sasiela WJ, Tamby JF, Tricoci P, White HD, Zeiher AM; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab and Cardiovascular Outcomes after Acute Coronary Syndrome. N Engl J Med. 2018 Nov 29;379(22):2097-2107. doi: 10.1056/NEJMoa1801174. Epub 2018 Nov 7. PMID 30403574
- [Background] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Background] Virani SS, Newby LK, Arnold SV, Bittner V, Brewer LC, Demeter SH, Dixon DL, Fearon WF, Hess B, Johnson HM, Kazi DS, Kolte D, Kumbhani DJ, LoFaso J, Mahtta D, Mark DB, Minissian M, Navar AM, Patel AR, Piano MR, Rodriguez F, Talbot AW, Taqueti VR, Thomas RJ, van Diepen S, Wiggins B, Williams MS; Peer Review Committee Members. 2023 AHA/ACC/ACCP/ASPC/NLA/PCNA Guideline for the Management of Patients With Chronic Coronary Disease: A Report of the American Heart Association/American College of Cardiology Joint Committee on Clinical Practice Guidelines. Circulation. 2023 Aug 29;148(9):e9-e119. doi: 10.1161/CIR.0000000000001168. Epub 2023 Jul 20. PMID 37471501
- [Background] Yang S, Hoshino M, Yonetsu T, Zhang J, Hwang D, Shin ES, Doh JH, Nam CW, Wang J, Chen S, Tanaka N, Matsuo H, Kubo T, Chang HJ, Kakuta T, Koo BK. Outcomes of non-ischaemic coronary lesions with high-risk plaque characteristics on coronary CT angiography. EuroIntervention. 2023 Jan 23;18(12):1011-1021. doi: 10.4244/EIJ-D-22-00562. PMID 36222756
- [Background] Lee JM, Choi KH, Koo BK, Park J, Kim J, Hwang D, Rhee TM, Kim HY, Jung HW, Kim KJ, Yoshiaki K, Shin ES, Doh JH, Chang HJ, Cho YK, Yoon HJ, Nam CW, Hur SH, Wang J, Chen S, Kuramitsu S, Tanaka N, Matsuo H, Akasaka T. Prognostic Implications of Plaque Characteristics and Stenosis Severity in Patients With Coronary Artery Disease. J Am Coll Cardiol. 2019 May 21;73(19):2413-2424. doi: 10.1016/j.jacc.2019.02.060. PMID 31097161
- [Background] Ferencik M, Mayrhofer T, Bittner DO, Emami H, Puchner SB, Lu MT, Meyersohn NM, Ivanov AV, Adami EC, Patel MR, Mark DB, Udelson JE, Lee KL, Douglas PS, Hoffmann U. Use of High-Risk Coronary Atherosclerotic Plaque Detection for Risk Stratification of Patients With Stable Chest Pain: A Secondary Analysis of the PROMISE Randomized Clinical Trial. JAMA Cardiol. 2018 Feb 1;3(2):144-152. doi: 10.1001/jamacardio.2017.4973. PMID 29322167
- [Background] Williams MC, Moss AJ, Dweck M, Adamson PD, Alam S, Hunter A, Shah ASV, Pawade T, Weir-McCall JR, Roditi G, van Beek EJR, Newby DE, Nicol ED. Coronary Artery Plaque Characteristics Associated With Adverse Outcomes in the SCOT-HEART Study. J Am Coll Cardiol. 2019 Jan 29;73(3):291-301. doi: 10.1016/j.jacc.2018.10.066. PMID 30678759
- [Background] SCOT-HEART Investigators; Newby DE, Adamson PD, Berry C, Boon NA, Dweck MR, Flather M, Forbes J, Hunter A, Lewis S, MacLean S, Mills NL, Norrie J, Roditi G, Shah ASV, Timmis AD, van Beek EJR, Williams MC. Coronary CT Angiography and 5-Year Risk of Myocardial Infarction. N Engl J Med. 2018 Sep 6;379(10):924-933. doi: 10.1056/NEJMoa1805971. Epub 2018 Aug 25. PMID 30145934
- [Background] Virmani R, Burke AP, Kolodgie FD, Farb A. Pathology of the thin-cap fibroatheroma: a type of vulnerable plaque. J Interv Cardiol. 2003 Jun;16(3):267-72. doi: 10.1034/j.1600-0854.2003.8042.x. PMID 12800406
- [Background] Koo BK, Hu X, Kang J, Zhang J, Jiang J, Hahn JY, Nam CW, Doh JH, Lee BK, Kim W, Huang J, Jiang F, Zhou H, Chen P, Tang L, Jiang W, Chen X, He W, Ahn SG, Yoon MH, Kim U, Lee JM, Hwang D, Ki YJ, Shin ES, Kim HS, Tahk SJ, Wang J; FLAVOUR Investigators. Fractional Flow Reserve or Intravascular Ultrasonography to Guide PCI. N Engl J Med. 2022 Sep 1;387(9):779-789. doi: 10.1056/NEJMoa2201546. PMID 36053504